CLINICAL TRIAL: NCT03213938
Title: Acupuncture for Chronic Prostatitis/Chronic Pelvic Pain Syndrome: a Multicenter Randomized Controlled Trial
Brief Title: Acupuncture for Chronic Prostatitis/Chronic Pelvic Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Liu Zhishun, Principal Investigator, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZZ10-012
Record Dates: First submitted 2017-07-05; First posted 2017-07-11 (Actual); Results first posted 2021-09-27 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Chronic Prostatitis With Chronic Pelvic Pain Syndrome
Keywords: Chronic prostatitis; chronic pelvic pain syndrome; acupuncture; randomized controlled trial
MeSH Terms: conditions — Prostatitis | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental): The participants in the acupuncture group will receive treatment that consists of 20 acupuncture sessions over an 8-week (3 sessions in each of the first 4 weeks, and 2 sessions in each of the remaining 4 weeks) period after baseline, each for 30 minutes. Hwato brand disposable acupuncture needles (size 0.30 × 75mm; size 0.30 × 40mm) will be used. Sanyinjiao (SP6), Zhongliao (BL33), Shenshu (BL23), and Huiyang (BL35), were selected as acupoints protocol. SP6 is on the tibial aspect of the leg, posterior to the medial border of the tibia, 3 cun superior to the prominence of the medial malleolus; BL32 is in the sacral region, in the second posterior sacral foramen; BL33 is in the third posterior sacral foramen; BL35 is in the buttock region, 0.5 cun lateral to the extremity of the coccyx.
  Interventions: Device: Acupuncture
- Sham acupuncture (Sham Comparator): The participants in the sham acupuncture group will receive shallow needling at bilateral sham BL23, BL33, BL35 and SP6. The protocol includes the same duration and frequency of sessions as for the acupuncture treatment, but the treatment was delivered superficially at non-acupuncture points 10-15 mm to the lateral of corresponding acupuncture and not above a meridian line (15mm to BL23, BL33 and BL35; 10mm to SP6). The Hwato brand disposable acupuncture needles (size 0.30 × 25mm) will be inserted with a depth of 2-3 mm without any manipulation.
  Interventions: Device: Sham acupuncture

INTERVENTIONS:
Device: Acupuncture — For acupuncture group, Hwato brand disposable acupuncture needles (size 0.30 × 75mm; size 0.30 × 40mm) will be used. Bilateral SP6, BL33, BL23, and BL35, were selected as acupoints protocol.
  Acupuncture group consists of 20 sessions over an 8-week period after baseline, each for 30 minutes, and will be administered over 8 weeks (3 sessions in each of the first 4 weeks, and 2 sessions in each of the remaining 4 weeks).
  Arms: Acupuncture
Device: Sham acupuncture — For sham acupuncture group, Hwato brand disposable acupuncture needles (size 0.30 × 25mm) will be used to insert vertically about 2-3 mm without manipulation into non-acupoints bilateral sham SP6, sham BL33, sham BL23, and sham BL35, which were located at different physical locations than SP6, BL23, BL 33, and BL35.
  Sham acupuncture group consists of 20 sessions over an 8-week period after baseline, each for 30 minutes, and will be administered over 8 weeks (3 sessions in each of the first 4 weeks, and 2 sessions in each of the remaining 4 weeks).
  Arms: Sham acupuncture

SUMMARY:
Chronic prostatitis/chronic pelvic pain syndrome (CP/CPPS) refers to the presence of bothersome pelvic pain symptoms without an identifiable cause. Common symptoms of CP/CPPS include discomfort in the perineum, suprapubic region, and lower urinary tract symptoms. It affects men of all ages without apparent racial predisposition, among which, 36-50 years old are the most commonly influenced. Yet, few effective therapies are available for treating CP/CPPS.

Acupuncture may be an effective treatment option for CP/CPPS. However, effects of acupuncture on CP/CPPS remain uncertain because of the small sample sizes or other methodological limitations.

The objective of this multi-centre, randomized, sham acupuncture-controlled trial is to assess the effectiveness of acupuncture for relieving symptoms of CP/CPPS. The results will provide a robust conclusion with a high level of evidence.

ELIGIBILITY:
Inclusion Criteria:

* 1.History of pain perceived in the prostate region and absence of other lower urinary tract pathology for a minimum of three of the past 6 months. In addition, any associated lower urinary tract symptoms, sexual function, and psychological factors should be addressed. Physical examinations, urinary analyses, and urine cultures will be performed for all subjects;
* 2. Age 18 to 50 years.
* 3. NIH Chronic Prostatitis Symptom Index (NIH- CPSI) total score ≥ 15.

Exclusion Criteria:

* 1. Prostate, bladder, or urethral cancer, seizure disorder in any medical history.
* 2. Inflammatory bowel disease, active urethral stricture, neurologic disease or disorder affecting the bladder, liver disease, neurologic impairment or psychiatric disorder preventing understanding of consent and self-report scale.
* 3. Urinary tract infection with a urine culture value of more than 100,000 CFU/mL, clinical evidence of urethritis, including urethral discharge or positive culture, diagnostic of sexually transmitted diseases (including gonorrhoea, chlamydia, mycoplasma or trichomonas, but not including HIV/AIDS), symptoms of acute or chronic epididymitis).
* 4. Residual urine volume≥100ML.
* 5. Qmax≤15ML/S.
* 6. Prior 4 weeks used androgen hormone inhibitors (finasteride), alpha-blockers (terazosin HCI, doxazosin mesylate, tamsulosin hydrochloride), antibiotics (ciprofloxacin hydrochloride), or any other prostatitis-specific medication (including herb and Chinese medicine).

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 440 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhishun Liu, Principal Investigator — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Guang'anmen Hospital, China Academy of Chinese Medical Science, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data and data dictionary will be available with publication until six months after publication.
  Formal request should be sent to the corresponding author (zhishunjournal@163.com) with a methodologically sound proposal.
  Researchers whose proposal has been approved will sign a data access agreement
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available with publication until until six months after publication.
Access Criteria: Formal request should be sent to the corresponding author (zhishunjournal@163.com) with a methodologically sound proposal. Researchers whose proposal has been approved.
  Researchers whose proposal has been approved will sign a data access agreement

REFERENCES:
- [Background] Qin Z, Liu Y, Zhou K, Wu J, Pang R, Li N, Xu C, Kwong JSW, Liu Z. Acupuncture for chronic prostatitis/chronic pelvic pain syndrome: study protocol for a randomized controlled trial. Trials. 2017 Dec 22;18(1):616. doi: 10.1186/s13063-017-2383-8. PMID 29273095
- [Result] Sun Y, Liu Y, Liu B, Zhou K, Yue Z, Zhang W, Fu W, Yang J, Li N, He L, Zang Z, Su T, Fang J, Ding Y, Qin Z, Song H, Hu H, Zhao H, Mo Q, Zhou J, Wu J, Liu X, Wang W, Pang R, Chen H, Wang X, Liu Z. Efficacy of Acupuncture for Chronic Prostatitis/Chronic Pelvic Pain Syndrome : A Randomized Trial. Ann Intern Med. 2021 Oct;174(10):1357-1366. doi: 10.7326/M21-1814. Epub 2021 Aug 17. PMID 34399062
- [Derived] Zhu L, Sun Y, Yan S, Liu X, Wang X, Liu Z. Efficacy of acupuncture on drinkers with chronic prostatitis / chronic pelvic pain syndrome: secondary analysis of a randomized clinical trial. Acupunct Med. 2024 Oct;42(5):243-250. doi: 10.1177/09645284241274158. Epub 2024 Sep 1. PMID 39219163
- [Derived] Zhu L, Fang J, Sun Y, Yang M, Yao H, Liu Z. Impact of ejaculation upon effect of acupuncture on chronic prostatitis/chronic pelvic pain syndrome: Secondary analysis of a randomized controlled trial. Integr Med Res. 2023 Jun;12(2):100943. doi: 10.1016/j.imr.2023.100943. Epub 2023 Apr 3. PMID 37122487

RESULTS

PARTICIPANT FLOW:
Groups:
- Acupuncture: The participants in the acupuncture group will receive treatment that consists of 20 acupuncture sessions over an 8-week (3 sessions in each of the first 4 weeks, and 2 sessions in each of the remaining 4 weeks) period after baseline, each for 30 minutes. Hwato brand disposable acupuncture needles (size 0.30 × 75mm; size 0.30 × 40mm) will be used. Sanyinjiao (SP6), Zhongliao (BL33), Shenshu (BL23), and Huiyang (BL35), were selected as acupoints protocol. SP6 is on the tibial aspect of the leg, posterior to the medial border of the tibia, 3 cun superior to the prominence of the medial malleolus; BL32 is in the sacral region, in the second posterior sacral foramen; BL33 is in the third posterior sacral foramen; BL35 is in the buttock region, 0.5 cun lateral to the extremity of the coccyx.
  Acupuncture: For acupuncture group, Hwato brand disposable acupuncture needles (size 0.30 × 75mm; size 0.30 × 40mm) will be used. Bilateral SP6, BL33, BL23, and BL35, were selected as acupoints protocol.
  Acupuncture group consists of 20 sessions over an 8-week period after baseline, each for 30 minutes, and will be administered over 8 weeks (3 sessions in each of the first 4 weeks, and 2 sessions in each of the remaining 4 weeks).
- Sham Acupuncture: The participants in the sham acupuncture group will receive shallow needling at bilateral sham BL23, BL33, BL35 and SP6. The protocol includes the same duration and frequency of sessions as for the acupuncture treatment, but the treatment was delivered superficially at non-acupuncture points 10-15 mm to the lateral of corresponding acupuncture and not above a meridian line (15mm to BL23, BL33 and BL35; 10mm to SP6). The Hwato brand disposable acupuncture needles (size 0.30 × 25mm) will be inserted with a depth of 2-3 mm without any manipulation.
  Sham acupuncture: For sham acupuncture group, Hwato brand disposable acupuncture needles (size 0.30 × 25mm) will be used to insert vertically about 2-3 mm without manipulation into non-acupoints bilateral sham SP6, sham BL33, sham BL23, and sham BL35, which were located at different physical locations than SP6, BL23, BL 33, and BL35.
  Sham acupuncture group consists of 20 sessions over an 8-week period after baseline, each for 30 minutes, and will be administered over 8 weeks (3 sessions in each of the first 4 weeks, and 2 sessions in each of the remaining 4 weeks).
Period: Overall Study
Arm/Group | Acupuncture | Sham Acupuncture
Started | 220 | 220
Completed | 206 | 208
Not Completed | 14 | 12
Not completed — Lost to Follow-up | 4 | 3
Not completed — Lack of Efficacy | 1 | 0
Not completed — Decline to participate | 5 | 4
Not completed — Without reason | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acupuncture | Sham Acupuncture | Total
Number analyzed (Participants) | 220 | 220 | 440
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (8.0) | 36.1 (7.9) | 35.8 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 220 | 220 | 440
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: 5 participants in the acupuncture and 4 participants in the sham acupuncture group declined to participate the trial.
  Participants
    Han: number analyzed (Participants) | 215 | 216 | 431
    Han | 213 | 214 | 427
    Others: number analyzed (Participants) | 215 | 216 | 431
    Others | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  China | 220 | 220 | 440
National Institutes of Health Chronic Prostatitis Symptom Index (NIH-CPSI) total score [Mean (Standard Deviation); unit: units on a scale] — The National Institutes of Health Chronic Prostatitis Symptom Index (NIH-CPSI) is a universally accepted, reliable and valid instrument recommended for clinical evaluation and research of CP/CPPS by consensus guidelines. It measures the domains of pain (score range, 0-21), urinary function (score range, 0-10) and quality of life impact (score range, 0-12) in CP/CPPS, with a total score ranging from 0 to 43 (a combination of subscale scores) and higher scores indicating worse conditions. Population: 5 participants in the acupuncture group declined to participate the trial and did not receive treatment.
  4 participants declined to participate the trial and 1 withdrew without reason in the sham acupuncture group. All those 5 participants did not receive treatment.
  units on a scale
    number analyzed (Participants) | 215 | 215 | 430
    (all) | 31.0 (4.8) | 31.4 (5.2) | 31.2 (5.0)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Responders at the End of 8-week
Description: The responder is defined as who has a decline of 6 or more than 6-point from baseline measured by using the National Institutes of Health Chronic Prostatitis Symptom Index (NIH-CPSI).
Time Frame: week 8
Measure: Number; unit: percentage of participants
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 220 | 220
percentage of participants | 60.6 | 36.8

2. Primary Outcome: Proportion of Responders at the End of 32-week
Description: The responder is defined as who has a decline of 6 or more than 6-point from baseline measured by using the NIH-CPSI.
Time Frame: week 32
Measure: Number; unit: percentage of participants
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 220 | 220
percentage of participants | 61.5 | 38.3

3. Secondary Outcome: Proportion of Responders at Other Time Points
Description: The responder is defined as who has a decline of 6 or more than 6-point from baseline measured by using the NIH-CPSI.
Time Frame: weeks 1-7; week 20
Measure: Number; unit: percentage of participants
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 220 | 220
percentage of participants
  Week 1 | 9.1 | 8.3
  Week 2 | 15.2 | 13.9
  Week 3 | 27.2 | 19.8
  Week 4 | 39.5 | 26.4
  Week 5 | 42.6 | 24.1
  Week 6 | 53.0 | 33.3
  Week 7 | 61.0 | 35.3
  Week 20 | 64.1 | 34.8

4. Secondary Outcome: the Change From Baseline in NIH-CPSI Total Score
Description: The National Institutes of Health Chronic Prostatitis Symptom Index (NIH-CPSI) is a universally accepted, reliable and valid instrument recommended for clinical evaluation and research of CP/CPPS by consensus guidelines. It measures the domains of pain (score range, 0-21), urinary function (0-10) and quality of life impact (0-12) in CP/CPPS, with a total score ranging from 0 to 43 and higher scores indicating worse conditions.
Time Frame: weeks 1-8; week 20; week 32
Population: Of the 220 participants randomly assigned to the acupuncture group, 206 completed 8-week treatment and 32-week follow-up: 5 declined to participate the trial, 4 lost to follow-up, 4 withdrew without reason and 1 withdrew because lack of perceived efficacy.
  Of the 220 participants randomly assigned to the sham acupuncture group, 208 completed 8-week treatment and 32-week follow-up: 4 declined to participate, 5 withdrew without reason and 3 lost to follow-up.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 215 | 214
score on a scale
  Week 1 | -1.9 [-2.4 to -1.5] | -1.3 [-1.8 to -0.9]
  Week 2: number analyzed (Participants) | 212 | 214
  Week 2 | -2.9 [-3.4 to -2.4] | -2.4 [-2.9 to -1.9]
  Week 3: number analyzed (Participants) | 210 | 214
  Week 3 | -3.9 [-4.4 to -3.4] | -3.0 [-3.5 to -2.5]
  Week 4: number analyzed (Participants) | 208 | 213
  Week 4 | -4.8 [-5.4 to -4.3] | -3.7 [-4.2 to -3.1]
  Week 5: number analyzed (Participants) | 207 | 211
  Week 5 | -5.2 [-5.8 to -4.6] | -3.7 [-4.3 to -3.2]
  Week 6: number analyzed (Participants) | 207 | 209
  Week 6 | -5.9 [-6.5 to -5.3] | -4.0 [-4.6 to -3.5]
  Week 7: number analyzed (Participants) | 206 | 208
  Week 7 | -6.7 [-7.3 to -6.1] | -4.6 [-5.2 to -4.0]
  Week 8: number analyzed (Participants) | 206 | 208
  Week 8 | -7.4 [-8.0 to -6.8] | -4.9 [-5.5 to -4.3]
  Week 20: number analyzed (Participants) | 206 | 208
  Week 20 | -7.2 [-8.0 to -6.6] | -4.5 [-5.2 to -3.9]
  Week 32: number analyzed (Participants) | 206 | 208
  Week 32 | -7.4 [-8.1 to -6.7] | -4.9 [-5.5 to -4.2]

5. Secondary Outcome: the Change From Baseline in NIH-CPSI Subscales
Description: The NIH-CPSI is a universally accepted, reliable and valid instrument recommended for clinical evaluation and research of CP/CPPS by consensus guidelines. It measures the domains of pain, urinary function and quality of life impact in CP/CPPS. The score range of pain subscale is 0-21, with higher scores indicating worse conditions. The score range of urinary function subscale is 0-10, with higher scores indicating worse conditions. The score range of quality-of-life subscale is 0-12, with higher scores indicating worse quality of life.
Time Frame: weeks 1-8; week 20; week 32
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 215 | 214
score on a scale
  Change in NIH-CPSI pain subscale at week 1 | -0.6 [-0.9 to -0.4] | -0.5 [-0.7 to -0.2]
  Change in NIH-CPSI pain subscale at week 2: number analyzed (Participants) | 212 | 214
  Change in NIH-CPSI pain subscale at week 2 | -0.8 [-1.1 to -0.6] | -0.8 [-1.0 to -0.5]
  Change in NIH-CPSI pain subscale at week 3: number analyzed (Participants) | 210 | 214
  Change in NIH-CPSI pain subscale at week 3 | -1.1 [-1.4 to -0.9] | -0.8 [-1.1 to -0.6]
  Change in NIH-CPSI pain subscale at week 4: number analyzed (Participants) | 208 | 213
  Change in NIH-CPSI pain subscale at week 4 | -1.6 [-1.8 to -1.3] | -1.1 [-1.3 to -0.9]
  Change in NIH-CPSI pain subscale at week 5: number analyzed (Participants) | 207 | 211
  Change in NIH-CPSI pain subscale at week 5 | -1.5 [-1.7 to -1.2] | -1.1 [-1.3 to -0.9]
  Change in NIH-CPSI pain subscale at week 6: number analyzed (Participants) | 207 | 209
  Change in NIH-CPSI pain subscale at week 6 | -1.8 [-2.0 to -1.5] | -1.1 [-1.4 to -0.9]
  Change in NIH-CPSI pain subscale at week 7: number analyzed (Participants) | 206 | 208
  Change in NIH-CPSI pain subscale at week 7 | -2.0 [-2.3 to -1.8] | -1.3 [-1.5 to -1.1]
  Change in NIH-CPSI pain subscale at week 8: number analyzed (Participants) | 206 | 208
  Change in NIH-CPSI pain subscale at week 8 | -2.1 [-2.4 to -1.9] | -1.3 [-1.5 to -1.1]
  Change in NIH-CPSI pain subscale at week 20: number analyzed (Participants) | 206 | 208
  Change in NIH-CPSI pain subscale at week 20 | -2.0 [-2.3 to -1.8] | -1.0 [-1.2 to -0.7]
  Change in NIH-CPSI pain subscale at week 32: number analyzed (Participants) | 206 | 208
  Change in NIH-CPSI pain subscale at week 32 | -2.0 [-2.3 to -1.8] | -1.3 [-1.5 to -1.0]
  Change in NIH-CPSI urinary subscale at week 1 | -0.5 [-0.7 to -0.3] | -0.4 [-0.6 to -0.2]
  Change in NIH-CPSI urinary subscale at week 2: number analyzed (Participants) | 212 | 214
  Change in NIH-CPSI urinary subscale at week 2 | -0.8 [-1.0 to -0.6] | -0.6 [-0.8 to -0.4]
  Change in NIH-CPSI urinary subscale at week 3: number analyzed (Participants) | 210 | 214
  Change in NIH-CPSI urinary subscale at week 3 | -1.0 [-1.3 to -0.8] | -0.9 [-1.1 to -0.7]
  Change in NIH-CPSI urinary subscale at week 4: number analyzed (Participants) | 208 | 213
  Change in NIH-CPSI urinary subscale at week 4 | -1.3 [-1.6 to -1.1] | -1.0 [-1.2 to -0.8]
  Change in NIH-CPSI urinary subscale at week 5: number analyzed (Participants) | 207 | 211
  Change in NIH-CPSI urinary subscale at week 5 | -1.6 [-1.8 to -1.3] | -1.1 [-1.3 to -0.9]
  Change in NIH-CPSI urinary subscale at week 6: number analyzed (Participants) | 207 | 209
  Change in NIH-CPSI urinary subscale at week 6 | -1.7 [-1.9 to -1.5] | -1.2 [-1.4 to -0.9]
  Change in NIH-CPSI urinary subscale at week 7: number analyzed (Participants) | 206 | 208
  Change in NIH-CPSI urinary subscale at week 7 | -1.9 [-2.2 to -1.7] | -1.3 [-1.6 to -1.1]
  Change in NIH-CPSI urinary subscale at week 8: number analyzed (Participants) | 206 | 208
  Change in NIH-CPSI urinary subscale at week 8 | -2.1 [-2.4 to -1.9] | -1.4 [-1.6 to -1.2]
  Change in NIH-CPSI urinary subscale at week 20: number analyzed (Participants) | 206 | 208
  Change in NIH-CPSI urinary subscale at week 20 | -2.1 [-2.3 to -1.8] | -1.5 [-1.7 to -1.2]
  Change in NIH-CPSI urinary subscale at week 32: number analyzed (Participants) | 206 | 208
  Change in NIH-CPSI urinary subscale at week 32 | -2.1 [-2.4 to -1.9] | -1.5 [-1.8 to -1.2]
  Change in NIH-CPSI quality of life subscale at week 1 | -0.8 [-0.9 to -0.6] | -0.5 [-0.7 to -0.3]
  Change in NIH-CPSI quality of life subscale at week 2: number analyzed (Participants) | 212 | 214
  Change in NIH-CPSI quality of life subscale at week 2 | -1.2 [-1.4 to -1.0] | -0.9 [-1.2 to -0.7]
  Change in NIH-CPSI quality of life subscale at week 3: number analyzed (Participants) | 210 | 214
  Change in NIH-CPSI quality of life subscale at week 3 | -1.7 [-1.9 to -1.5] | -1.2 [-1.4 to -1.0]
  Change in NIH-CPSI quality of life subscale at week 4: number analyzed (Participants) | 208 | 213
  Change in NIH-CPSI quality of life subscale at week 4 | -1.9 [-2.2 to -1.7] | -1.5 [-1.8 to -1.3]
  Change in NIH-CPSI quality of life subscale at week 5: number analyzed (Participants) | 207 | 211
  Change in NIH-CPSI quality of life subscale at week 5 | -2.2 [-2.4 to -1.9] | -1.5 [-1.8 to -1.3]
  Change in NIH-CPSI quality of life subscale at week 6: number analyzed (Participants) | 207 | 209
  Change in NIH-CPSI quality of life subscale at week 6 | -2.4 [-2.7 to -2.2] | -1.7 [-2.0 to -1.5]
  Change in NIH-CPSI quality of life subscale at week 7: number analyzed (Participants) | 206 | 208
  Change in NIH-CPSI quality of life subscale at week 7 | -2.8 [-3.0 to -2.5] | -1.9 [-2.2 to -1.7]
  Change in NIH-CPSI quality of life subscale at week 8: number analyzed (Participants) | 206 | 208
  Change in NIH-CPSI quality of life subscale at week 8 | -3.1 [-3.4 to -2.8] | -2.2 [-2.4 to -1.9]
  Change in NIH-CPSI quality of life subscale at week 20: number analyzed (Participants) | 206 | 208
  Change in NIH-CPSI quality of life subscale at week 20 | -3.2 [-3.5 to -2.8] | -2.0 [-2.4 to -1.7]
  Change in NIH-CPSI quality of life subscale at week 32: number analyzed (Participants) | 206 | 208
  Change in NIH-CPSI quality of life subscale at week 32 | -3.1 [-3.5 to -2.8] | -2.1 [-2.4 to -1.8]

6. Secondary Outcome: the Change From Baseline in the International Prostate Symptom Score (IPSS)
Description: IPSS is a valid, reliable and sensitive measure for patients with lower urinary tract symptoms; it is widely used in clinical practice and research to determine the severity of lower urinary tract symptoms, including incomplete bladder emptying, frequency of urination, intermittency, urgency, weak urine stream, straining and nocturia. Each of the questions is rated from 0 (not at all) to 5 (almost always). IPSS score ranges from 0 to 35, with higher score indicating more severe urinary symptoms.
Time Frame: week 4; week 8; week 20; week 32
Population: Of the 220 participants randomly assigned to the acupuncture group, 206 completed 8-week treatment and 32-week follow-up. Additionally, the data of IPSS was not available for one participant at week 32 in the acupuncture group.
  Of the 220 participants randomly assigned to the sham acupuncture group, 208 completed 8-week treatment and 32-week follow-up.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 208 | 213
score on a scale
  Week 4 | -2.7 [-3.2 to -2.3] | -1.7 [-2.1 to -1.2]
  Week 8: number analyzed (Participants) | 206 | 208
  Week 8 | -4.4 [-4.9 to -3.9] | -2.7 [-3.2 to -2.2]
  Week 20: number analyzed (Participants) | 206 | 208
  Week 20 | -4.7 [-5.3 to -4.2] | -3.0 [-3.6 to -2.4]
  Week 32: number analyzed (Participants) | 205 | 208
  Week 32 | -4.7 [-5.4 to -4.1] | -3.1 [-3.8 to -2.5]

7. Secondary Outcome: the Change From Baseline in the Hospital Anxiety and Depression Scale (HADS)
Description: HADS is made up of 7 items for the assessment of depression and anxiety; the completion of this scale usually requires 2-5 minutes. HADS score ranges from 0 to 42, with higher scores indicating greater anxiety and depression.
Time Frame: week 8; week 20; week 32
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 206 | 208
score on a scale
  Week 8 | -1.9 [-2.5 to -1.4] | -0.8 [-1.3 to -0.3]
  Week 20 | -2.4 [-3.0 to -1.8] | -0.6 [-1.3 to 0.0]
  Week 32 | -2.8 [-3.5 to -2.2] | -0.5 [-1.2 to 0.1]

8. Secondary Outcome: the Change From Baseline in the International Index of Erectile Function 5 (IIEF-5)
Description: The IIEF-5 is a psychometrically valid and reliable instrument with high sensitivity and specificity for detecting treatment effects in patients with erection dysfunction of a broad spectrum of aetiology. Chinese version IIEF-5 score ranges from 0 to 25, with lower scores indicating greater severity of dysfunction and minimal clinical important difference over 5.
Time Frame: week 8; week 20; week 32
Population: Of the 220 participants randomly assigned to the acupuncture group, 206 completed 8-week treatment and 32-week follow-up. Additionally, the data of IIEF-5 was not available for two participants at week 32.
  Of the 220 participants randomly assigned to the sham acupuncture group, 208 completed 8-week treatment and 32-week follow-up. Additionally, the data of IIEF-5 was not available for one participant at weeks 8, 20 and 32.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 206 | 207
score on a scale
  Week 8 | 0.8 [0.2 to 1.3] | 0.3 [-0.3 to 0.8]
  Week 20 | 0.7 [0.2 to 1.3] | 0.2 [-0.3 to 0.7]
  Week 32: number analyzed (Participants) | 204 | 207
  Week 32 | 1.0 [0.4 to 1.6] | 0.4 [-0.1 to 1.0]

9. Secondary Outcome: the Change From Baseline in the European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L) Questionnaire
Description: The EQ-5D-5L is a well-established and suitable for evaluation of quality of life in participants with CP/CPPS. EQ-5D-5L overall index ranges from -0.39 to 1.00, with higher overall index indicating better generic health-status.
Time Frame: week 8; week 20; week 32
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 206 | 208
units on a scale
  Week 8 | 0.06 [0.05 to 0.07] | 0.03 [0.02 to 0.04]
  Week 20 | 0.06 [0.05 to 0.07] | 0.03 [0.02 to 0.04]
  Week 32 | 0.06 [0.05 to 0.08] | 0.03 [0.02 to 0.04]

10. Secondary Outcome: the Proportions of Participants in Each Response Category of the Global Response Assessment (GRA)
Description: GRA consists of 7 response categories: markedly worsened, moderately worsened, slightly worsened, no change, slightly improved, moderately improved, and markedly improved.
Time Frame: week 4; week 8; week 20; week 32
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 208 | 213
percentage of participants
  Week 4 : Markedly improved | 15.9 | 7.5
  Week 4 : Moderately improved | 24.0 | 14.6
  Week 4 : Slightly improved | 46.6 | 50.7
  Week 4 : No change | 13.0 | 25.4
  Week 4 : Slightly worsened | 0.5 | 1.9
  Week 4 : Moderately worsened | 0 | 0
  Week 4 : Markedly worsened | 0 | 0
  Week 8 : Markedly improved: number analyzed (Participants) | 206 | 208
  Week 8 : Markedly improved | 30.6 | 8.7
  Week 8 : Moderately improved | 36.4 | 27.9
  Week 8 : Slightly improved | 27.2 | 40.9
  Week 8 : No change | 5.3 | 19.2
  Week 8 : Slightly worsened | 0.5 | 3.4
  Week 8 : Moderately worsened | 0 | 0
  Week 8 : Markedly worsened | 0 | 0
  Week 20 : Markedly improved: number analyzed (Participants) | 206 | 208
  Week 20 : Markedly improved | 24.3 | 6.7
  Week 20 : Moderately improved | 24.3 | 17.8
  Week 20 : Slightly improved | 27.7 | 31.7
  Week 20 : No change | 19.4 | 30.3
  Week 20 : Slightly worsened | 4.4 | 12.0
  Week 20 : Moderately worsened | 0 | 1.4
  Week 20 : Markedly worsened | 0 | 0
  Week 32 : Markedly improved: number analyzed (Participants) | 206 | 208
  Week 32 : Markedly improved | 22.3 | 8.2
  Week 32 : Moderately improved | 24.8 | 16.8
  Week 32 : Slightly improved | 27.2 | 29.3
  Week 32 : No change | 20.9 | 32.7
  Week 32 : Slightly worsened | 4.4 | 8.7
  Week 32 : Moderately worsened | 0.5 | 3.9
  Week 32 : Markedly worsened | 0 | 0.5

11. Secondary Outcome: the Change for Peak and Average Urinary Flow Rate From Baseline
Time Frame: weeks 8 and 32
Population: Of the 220 participants randomly assigned to the acupuncture group, 206 completed 8-week treatment and 32-week follow-up.
  Of the 220 participants randomly assigned to the sham acupuncture group, 208 completed 8-week treatment and 32-week follow-up.
  Additionally, the data of peak and average urinary flow rate was not available for several participants.
Measure: Mean (95% Confidence Interval); unit: ml/s
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 195 | 198
ml/s
  Changes in peak urinary flow rate at week 8 | 0.6 [-0.3 to 1.6] | 0.7 [-0.2 to 1.6]
  Changes in peak urinary flow rate at week 32: number analyzed (Participants) | 186 | 187
  Changes in peak urinary flow rate at week 32 | 0.5 [-0.4 to 1.3] | -0.6 [-1.4 to 0.2]
  Changes in average urinary flow rate at week 8: number analyzed (Participants) | 195 | 195
  Changes in average urinary flow rate at week 8 | 0.6 [0.1 to 1.1] | 0.4 [-0.1 to 0.9]
  Changes in average urinary flow rate at week 32: number analyzed (Participants) | 186 | 187
  Changes in average urinary flow rate at week 32 | 0.5 [0.1 to 1.0] | -0.2 [-0.6 to 0.3]

12. Other Pre Specified Outcome: Expectation Assessment
Description: Expectation assessment will be assessed at baseline, which includes 2 brief questions to investigate whether patients are confident that acupuncture treatment will help their CP/CPPS: "In general, is acupuncture effective for controlling the illness?", "Do you think acupuncture will helpful to improve your CP/CPPS symptoms?" For each question, participants could choose "Yes", "No" or "unclear" as the answer.
Time Frame: baseline
Population: 5 participants in the acupuncture group declined to participate the trial and did not receive treatment. Additionally, the data of expectation assessment was not available for 2 participants in the acupuncture group.
  4 participants declined to participate the trial and 1 withdrew without reason in the sham acupuncture group. All those 5 participants did not receive treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 213 | 215
Participants
  Do you believe acupuncture is effective for treating diseases in general?: Yes | 167 | 165
  Do you believe acupuncture is effective for treating diseases in general?: No | 0 | 1
  Do you believe acupuncture is effective for treating diseases in general?: Unclear | 46 | 49
  Do you think acupuncture will be helpful to improve your CP/CPPS symptoms?: Yes | 156 | 150
  Do you think acupuncture will be helpful to improve your CP/CPPS symptoms?: No | 0 | 1
  Do you think acupuncture will be helpful to improve your CP/CPPS symptoms?: Unclear | 57 | 64

ADVERSE EVENTS:
Time Frame: 34 weeks
Arm/Group | Acupuncture | Sham Acupuncture
All-Cause Mortality (participants affected / at risk) | 0/220 | 0/220
Serious Adverse Events (participants affected / at risk) | 0/220 | 0/220
Other Adverse Events (participants affected / at risk) | 20/220 | 14/220
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Acupuncture (N=220) | Sham Acupuncture (N=220)
Subcutaneous hematoma (Skin and subcutaneous tissue disorders) | 9 | 5
Localized infection (Infections and infestations) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Cold (General disorders) | 7 | 6
Fever (General disorders) | 1 | 1
Tonsillitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute gastritis (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-09-04): https://cdn.clinicaltrials.gov/large-docs/38/NCT03213938/Prot_SAP_ICF_000.pdf